CLINICAL TRIAL: NCT04913142
Title: About Oral and Gut Microbiota in Intensive Care Unit : SARS-CoV-2 (COVID-19) Infection Impact. (CO-MIC Study)
Brief Title: About Oral and Gut Microbiota in Intensive Care Unit : SARS-CoV-2 (COVID-19) Infection Impact.
Acronym: CO-MIC
Status: Withdrawn | Type: Observational
Why Stopped: No more COVID+ patients to enrolled
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/21/0019; 2021-A00096-35 (Other: ID-RCB)
Record Dates: First submitted 2021-05-31; First posted 2021-06-04 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: SARS-CoV-2 Acute Respiratory Disease
Keywords: SARS-CoV-2; COVID 19; Critical care; microbiota; microbiome
MeSH Terms: conditions — COVID-19 | interventions — Defecation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fecal and oral samples will be collected in each patient at the admission in intensive care unit to analyze bacterial DNA and describe their microbiota
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control: patients not suffering from COVID-19 hospitalized in intensive care unit
  Interventions: Other: Fecal and oral samples
- patients COVID-19: patients suffering from COVID-19 hospitalized in intensive care unit
  Interventions: Other: Fecal and oral samples

INTERVENTIONS:
Other: Fecal and oral samples — oral and rectal swab from patients hospitalized at day 1, each 7 days and at the end of their ICU stay

SUMMARY:
The objective of the present study is to describe the negative impact on oral and gut microbiota of a severe acute respiratory syndrome SARS-CoV-2 infection in patients hospitalized in intensive care units (ICU). The study would like to compare their microbiota to the microbiota of ICU patients, non-infected by the SARS-CoV-2.

DETAILED DESCRIPTION:
Gut microbiota in ICU patients is sorely distorted, there is an important loss of diversity which can be traduced by a decrease of commensal bacteria and an increase of pathogens. The virulence, infectivity, and transmissibility of the emerging SARS-Coronavirus 2 is a reason for us to find strategies and therapeutics to curb the epidemic. Gut mucosa is very probably a target for the virus and it seems likely that feces are a way of transmissibility. It suppose too that gut microbiota is more weathered in patients with a SARS-CoV-2 infection, moreover if they have to be hospitalized in ICU. For this reason, the present study would like to collect oral and rectal swab from patients hospitalized in ICU for a serious SARS-CoV-2 infection and from patients hospitalized in ICU for another reason that a SARS-CoV-2 infection at day 1, each 7 days and at the end of their ICU stay. Other objectives are to know if this distorted microbiota is a risk factor for poor outcomes in our ICU patients, if antibiotics and artificial nutrition are too a risk factor of weathered microbiota and finally if we can connect oral and rectal dysbiosis to use the oral dysbiosis to predict the rectal dysbiosis in view of the ease to collect oral sample.

ELIGIBILITY:
Inclusion Criteria:

Controls:

- Hospitalized patient with non-SARS-CoV-2 hypoxemic pneumonia

Patients COVID 19:

- Patient hospitalized for SARS-CoV-2 hypoxemic pneumonia

All:

* Patient hospitalized for less than 48 hours in a general intensive care unit
* Patient who has given free, informed and express (oral) consent to participate in the research (or a close relative or trusted person of the patient if the patient cannot express himself/herself)
* Patient covered by a social security system or equivalent
* Expected hospitalization of more than 48 hours

Exclusion Criteria:

* gut inflammatory disease
* recent gut surger
* ostomy
* recent antibiotics
* artificial nutrition in the long term

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients hospitalized in intensive care units (ICU)
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Constitution of the oral and faecal microbiota obtained by sequencing of bacterial DNA | day 1
  measuring the difference in bacterial DNA sequencing from oral and fecal samples among ICU patients infected by the SARS-CoV-2 and ICU patients without SARS-CoV-2 at day 1
Measuring the difference in bacterial DNA sequencing from oral and fecal samples of patients infected by the SARS-COV-2 and patient without SARS-COV-2 at day 7 | day 7
  Measuring difference in bacterial DNA sequencing from oral and fecal samples among ICU patients infected by the SARS-CoV-2 and ICU patients without SARS-CoV-2
Measuring the difference in bacterial DNA sequencing from oral and fecal samples of patient infected by the SARS-COV-2 and patient without SARS-COV-2 at day 14 | day 14
  difference in bacterial DNA sequencing from oral and fecal samples among ICU patients infected by the SARS-CoV-2 and ICU patients without SARS-CoV-2

CONTACTS AND LOCATIONS:
Overall Officials: Fanny BOUNES, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No